CLINICAL TRIAL: NCT02489617
Title: The Incidence of Adjacent Synchronous Ipsilateral Infiltrating Carcinoma and/or DCIS in Patients Diagnosed With Intraductal Papilloma Without Atypia or Flat Epithelial Atypia by Core Needle Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Faina Nakhlis, MD, Faina Nakhlis, MD, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-174
Record Dates: First submitted 2015-06-18; First posted 2015-07-03 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Flat Epithelia Atypia; Intraductal Papilloma Without Atypia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (1):
- Pathologic evaluation of excised tissue (Experimental): Patient diagnosed with intraductal papilloma without atypia (IPWA) or flat epithelial atypia (FEA).
  -- Pathologic evaluation of excised tissue
  Interventions: Other: Pathologic evaluation of excised tissue

INTERVENTIONS:
Other: Pathologic evaluation of excised tissue — Up to 3 months after excisional biopsy

SUMMARY:
This research study is studying a surgical intervention to rule out the presence of cancer in participants that have been diagnosed with flat epithelial atypia (FEA) or intraductal papilloma without atypia (IPWA) by core needle biopsy.

DETAILED DESCRIPTION:
Breast milk is made in lobules and is carried through the ducts toward the nipple. Normal ducts are lined by one layer of cells very similar to each other in appearance. Flat epithelia atypia (FEA) and intraductal papilloma without atypia (IPWA) are changes seen within the milk ducts. In the recent years these lesions have been seen more often, seemingly because more core needle biopsies are being done with the help of a mammogram, ultrasound or breast MRI. The reason for this is there is new technology available which is able to do such biopsies. A core needle biopsy uses a hollow needle to remove samples of tissue from the breast. This is an accurate method that does not involve surgery.

FEA and IPWA are not very common and there are few research studies addressing them. Women found to have FEA or IPWA on core biopsy results may receive conflicting recommendations about how to precede next. It is unclear if more tissue should be removed from the biopsy site to ensure that there is no cancer nearby.

The purpose of this study is to find out how often cancer is identified by excisional biopsy near an initial core biopsy where FEA or IPWA has previously been seen. Depending on these findings doctors will be better able to advise their patients as to whether they need to have a surgical biopsy, when FEA or IPWA are seen on needle biopsy, to rule out the presence of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women all races and ethnic groups are eligible for this trial. This trial is open to the accrual of women only.
* Patients must be women
* Patients must be at least 18 years of age
* Patients must have an imaging abnormality that necessitated a core needle biopsy
* The imaging abnormality must have been categorized as Breast Imaging-Reporting and Data System (BIRADS) level 1-4 lesion
* There is documented concordance* between the initial breast imaging finding and the core biopsy pathology report. The core needle biopsy must contain FEA or IPWA, according to the local pathologist. (It is possible that the central pathology review which is done after the patient is registered on this protocol will have a diagnosis discrepant from that made by the original institution's pathologist. In that case, the study team will communicate this to the original institution's site investigator within one week of the date of the central pathology review having been finalized). Patients may have a personal history of prior or concurrent fibroadenoma and a prior history of proliferative breast lesions with or without atypia.
* Patients must be registered on study within 100 days after core needle biopsy.
* Patients must have an ability to understand and the willingness to sign a written informed consent document. The patient is still eligible for this study even if she declines consent for her tissue to be used for any (or all) of the correlative studies described in this document and/or if she declines consent for her tissue to go into a tissue bank for future unspecified research.

  * Concordance is a determination by the radiologist (or his or her covering provider) performing an image-guided core needle biopsy that the pathology report from this procedure corresponds to the imaging appearance of a given lesion and that the said lesion's most representative portion has been sampled.

Exclusion Criteria:

* Personal history and/or concomitant diagnosis of invasive breast cancer or DCIS
* Palpable abnormality diagnosed by core needle biopsy to be FEA or IPWA
* Pathologic nipple discharge associated with IPWA (spontaneous bloody or clear persistent single duct discharge)
* A BIRADS 5 lesion
* Discordance between the initial breast imaging finding and the core biopsy pathology report
* The presence of atypical ductal hyperplasia (ADH) on core biopsy
* Known current pregnancy. A pregnancy test is not required for this exclusion criteria.
* Women who are breastfeeding
* Patient registered on study more than 100 days since the date of core needle biopsy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2025-06 (Actual)

PRIMARY OUTCOMES:
Rate of invasive carcinoma and/or DCIS in patients originally diagnosed with FEA or IPWA on core biopsy, based on local pathology review | 60 days

SECONDARY OUTCOMES:
Rate of invasive carcinoma and/or DCIS in patients originally diagnosed with FEA or IPWA on core biopsy, based on central pathology review | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Faina Nakhlis, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (18):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Georgetown University, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Indiana University, Indianapolis, Indiana
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - MedStar Franklin Square Medical Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Howard County General Hospital, Columbia, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial SLoan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - University of North Carolina - Hillsborough Campus, Hillsborough, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided